CLINICAL TRIAL: NCT04663035
Title: CT-guided Thermal Ablation Plus Tislelizumab Versus Ablation Alone for Intrahepatic Recurrent Early Stage Hepatocellular Carcinoma: a Randomized Controlled Phase II Clinical Trial
Brief Title: Ablation Plus Tislelizumab Versus Ablation Alone for Intrahepatic Recurrent Early Stage HCC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ming Zhao (Other)
Responsible Party: Sponsor-Investigator, Ming Zhao, Professor, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2020-195-01
Record Dates: First submitted 2020-12-09; First posted 2020-12-10 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Recurrent Hepatocellular Carcinoma
Keywords: Recurrent Hepatocellular Carcinoma; Ablation; Tislelizumab
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ablation Plus Tislelizumab (Experimental): Patients in this arm will receive ablation followed by tislelizumab, which will be started within 3-7 days after ablation until disease progression or intolerable toxicity, for 12 months.
  Interventions: Drug: Tislelizumab; Procedure: Ablation
- Ablation Alone (Active Comparator): Patients in this group will receive ablation therapy and then enter the follow-up phase.
  Interventions: Procedure: Ablation

INTERVENTIONS:
Drug: Tislelizumab — 200mg, iv. drip, Q3W. Tislelizumab will start within 3-7 days after ablation treatment. The longest course of treatment is 12 months.
  Other Names: Tislelizumab Injection
  Arms: Ablation Plus Tislelizumab
Procedure: Ablation — After local anesthesia and intravenous sedative injection, the unipolar needle would be gradually inserted into the lesion and placed on the deepest edge of the lesion. The ablation electrode is a unipolar needle with a bare end of 2 or 3 cm (adjusted to tumor size). The ablation power is 150 watts (range from 100 to 200 watts). In general, the average ablation time for each lesion is about 12 minutes (ranging from 10 to 15 minutes).

SUMMARY:
This is a randomized, controlled, phase 2 study to assess the efficacy and safety of ablation followed by tislelizumab versus ablation alone in patients with early recurrent hepatocellular carcinoma.

DETAILED DESCRIPTION:
Ablation is one of the main treatments for early recurrent HCC, and its immune stimulation is expected to improve the efficacy of anti-PD-1 immune checkpoint inhibitor therapy. Tislelizumab is a new immunotherapy agent with independent intellectual property rights in China, which is highly efficient and safe. It is of great value to combine Tislelizumab with ablation to reduce the risk of recurrence in HCC patients. In this study, early-stage HCC patients with high risk of recurrence would be included and randomly assigned to receive ablation plus Tislelizumab or ablation alone. The tumor recurrence, overall survival and safety would be observed and recorded to analyze whether Tislelizumab can reduce the recurrence rate.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological diagnosed HCC.
2. The recurrent lesions should meet the diagnostic and staging criteria of the Barcelona liver cancer clinical system (BCLC) recommended by the American Association of liver Diseases and the European Association of liver Diseases (AASLD/EASL). The specific diagnostic criteria for HCC are as follows:

   I. Intrahepatic lesions ≥ 1cm, with typical HCC findings in dynamic contrast-enhanced CT or MRI, that is, enhancement in arterial phase or decreased enhancement in portal phase.

   II. Intrahepatic lesions ≥ 1cm without typical imaging findings, the biopsy can be performed.

   III. Intrahepatic lesions < 1cm, ultrasound follow-up every 4 months, if the enlargement exceeds 1cm, then refer to standard I or II.
3. If the intrahepatic recurrent lesions are diagnosed by the above criteria, BCLC-0/A stage can be performed as follows:

   I. BCLC-0: single lesion < 2cm, Child-Pugh A (without ascites), and ECOG-PS 0. II.BCLC-A: single lesion ≥ 2cm, Child-Pugh A (without ascites), and ECOG-PS 0. III.BCLC-A stage: 2-3 lesions but all are less than 3cm. Child-Pugh A (without ascites), and ECOG-PS 0.
4. The recurrence time of HCC should be between 3 and 12 months.
5. Patients with recurrent HCC lesions should meet the indications of ablation treatment, as follows:

I. Single lesion ≤ 5 cm; or. II. 2-3 lesions, all are less than 3cm; and. III. The location of the above lesions should be far away from the dangerous sites.

6. Life expectancy ≥ 12 months. 7. The laboratory test shall be completed within 7 days before the screening and the following criteria shall be met: I. Adequate hematologic function：

1. WBC ≥ 2.0 x 109/L (stable, off any growth factor within 4 weeks of study drug administration)
2. Neutrophils ≥ 1.5 x 109/L (stable, off any growth factor within 4 weeks of study drug administration)
3. Platelets ≥ 60 x 109/L (transfusion to achieve this level is not permitted)
4. Hemoglobin ≥ 80 g/L (may be transfused to meet this requirement)

II. Adequate hepatic function:

1. Serum Aspartate Aminotransferase (AST) < 8 X ULN
2. Serum Alanine Aminotransferase (ALT) < 8 X ULN
3. Serum total bilirubin < 3 mg/dL
4. Serum albumin ≥ 2.8 g/dL

III. Adequate coagulation function:

a)Prothrombin time (PT)-international normalized ratio (INR)≤ 2.3 or PT < 6 seconds above control

IV. Adequate renal function:

1. Creatinine Crack >40 mL/min (Cockcroft-Gault formula) a serum creatinine of < 1.5 × ULN

   Exclusion Criteria:

   -Target lesion

   1. Known fibrolamellar HCC, sarcomatous HCC, or mixed cholangiocarcinoma and HCC.

   2. Patients who have undergone a liver transplant or those who are in the waiting list for liver transplantation.

   3. With vascular invasion and extrahepatic metastases.
   * General condition

     1. Patients with cardiac pacemaker implantation. 2. Any history of hepatic encephalopathy. 3. Any prior (within 1 year) or current clinically significant ascites as measured by physical examination and that requires active paracentesis for control.

     4. Any history of clinically meaningful variceal bleeding within the last 3 months 5. Hepatitis B virus DNA copy number > 500 IU/mL. 6. Hepatitis D infection in subjects with hepatitis B. 7. Prior malignancy active within the previous 5 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, prostate cancer without evidence of PSA progression or carcinoma in situ such as the following: gastric, prostate, cervix, colon, melanoma, or breast for example.

     8. Subjects with any active autoimmune disease or history of known or suspected autoimmune disease except for subjects with vitiligo, resolved childhood asthma/atopy, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.

     9. Uncontrolled or clinically significant cardiac disease. 10. Positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
   * Previous / concomitant therapy

     1. Prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti- CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
     2. Prior organ allograft or allogeneic bone marrow transplantation
     3. All toxicities attributed to prior anti-cancer therapy other than neuropathy, alopecia and fatigue must have resolved to Grade 1 (NCI CTCAE version 5.0) or baseline before administration of study drug. Subjects with toxicities attributed to prior anti-cancer therapy which are not expected to resolve and result in long lasting sequelae are permitted to enroll. Neuropathy must have resolved to Grade 2 (NCI CTCAE version 5.0).
     4. Active bacterial or fungal infections requiring systemic treatment within 7 days
     5. Use of other investigational drugs (drugs not marketed for any indication) within 28 days or at least 5 half-lives (whichever is longer) before study drug administration
     6. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses > 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-21 (Actual); Primary Completion 2023-12-18 (Estimated); Study Completion 2025-12-18 (Estimated)

PRIMARY OUTCOMES:
1-year recurrence-free survival (RFS) rate | 1 year
  It is defined as the percentage of patients who achieve a time interval of 1 year of no disease recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (by any cause) from date of enrollment, whichever occurs first.

SECONDARY OUTCOMES:
2-year recurrence-free survival (RFS) rate | 2 years
  It is defined as the percentage of patients who achieve a time interval of 2 year of no disease recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (by any cause) from date of enrollment.
3-year recurrence-free survival (RFS) rate | 3 years
  It is defined as the percentage of patients who achieve a time interval of 3 year of no disease recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis) or death (by any cause) from date of enrollment.
Overall survival (OS) | 3 years
  It is defined as the time from date of randomization to the date of death (due to any cause). Subjects who are alive will be censored at the last known alive dates.
Time to Recurrence (TTR) | From date of randomization up to 5 years, approximately
  It is defined as the time between the date of enrollment and the date of first recurrence (i.e., intrahepatic recurrence or extrahepatic metastasis).
Safety of ablation and ablation plus Tislelizumab | From date of randomization up to 5 years, approximately
  Incidence of adverse events (AEs), serious AEs, deaths and laboratory abnormalities in all treated patients.
Biomarkers in tumor and peripheral blood to evaluate association with clinical efficacy and/or incidence of AEs. | From date of randomization up to 5 years, approximately
  Correlation of selected biomarkers with efficacy (RFS rate and OS) and safety (incidence of AEs) endpoints.
Evaluate the patient's cancer-related QoL using the European Organization for Research and Treatment of Cancer (EORTC) QOL questionnaire (QLQ), the EORTC QLQ-C30 and the EORTC QLQ-HCC18. | From date of randomization up to 5 years, approximately
  Change in sub-scale and total scores of EORTC QLQ-C30 and EORTC QLQ- HCC18 from baseline through follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Zhao, MD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Department of Minimally Invasive and Interventional Radiology, Liver Cancer Study and Service Group, Sun Yat-sen University Cancer Center,, Guangzhou, Guangdong, China

REFERENCES:
- [Background] Lyu N, Kong Y, Li X, Mu L, Deng H, Chen H, He M, Lai J, Li J, Tang H, Lin Y, Zhao M. Ablation Reboots the Response in Advanced Hepatocellular Carcinoma With Stable or Atypical Response During PD-1 Therapy: A Proof-of-Concept Study. Front Oncol. 2020 Oct 9;10:580241. doi: 10.3389/fonc.2020.580241. eCollection 2020. PMID 33163408
- [Background] Pan T, Xie QK, Lv N, Li XS, Mu LW, Wu PH, Zhao M. Percutaneous CT-guided Radiofrequency Ablation for Lymph Node Oligometastases from Hepatocellular Carcinoma: A Propensity Score-matching Analysis. Radiology. 2017 Jan;282(1):259-270. doi: 10.1148/radiol.2016151807. Epub 2016 Jul 11. PMID 27399327
- [Background] Deng H, Kan A, Lyu N, Mu L, Han Y, Liu L, Zhang Y, Duan Y, Liao S, Li S, Xie Q, Gao T, Li Y, Zhang Z, Zhao M. Dual Vascular Endothelial Growth Factor Receptor and Fibroblast Growth Factor Receptor Inhibition Elicits Antitumor Immunity and Enhances Programmed Cell Death-1 Checkpoint Blockade in Hepatocellular Carcinoma. Liver Cancer. 2020 Jun;9(3):338-357. doi: 10.1159/000505695. Epub 2020 Feb 25. PMID 32647635
- [Background] Lyu N, Kong Y, Pan T, Mu L, Sun X, Li S, Deng H, Lai J, Zhao M. Survival benefits of computed tomography-guided thermal ablation for adrenal metastases from hepatocellular carcinoma. Int J Hyperthermia. 2019;36(1):1003-1011. doi: 10.1080/02656736.2019.1663279. PMID 31544545
- [Background] Mu L, Pan T, Lyu N, Sun L, Li S, Xie Q, Deng H, Wu P, Liu H, Zhao M. CT-guided percutaneous radiofrequency ablation for lung neoplasms adjacent to the pericardium. Lung Cancer. 2018 Aug;122:25-31. doi: 10.1016/j.lungcan.2018.05.004. Epub 2018 May 12. PMID 30032841